CLINICAL TRIAL: NCT04992195
Title: Impact of COVID-19 Vaccines on Cerebrovascular Health - a Population-based Study
Brief Title: Impact of COVID-19 Vaccines on Cerebrovascular Health
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. IP Yiu Ming Bonaventure, Clinical Lecturer, Chinese University of Hong Kong
Other Study IDs: CREC No. 2021.386
Record Dates: First submitted 2021-08-03; First posted 2021-08-05 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Stroke, Acute; Stroke, Ischemic; Dementia; Brain Ischemia; Alzheimer Disease; Brain Diseases; Major Adverse Cardiovascular Event; Arterial Thromboembolism; Venous Thromboembolism
MeSH Terms: conditions — Stroke; Ischemic Stroke; Dementia; Brain Ischemia; Alzheimer Disease; Brain Diseases; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccination Group: Citizens who received baseline cognitive assessment and evaluation of metabolic risk factors from the CUHK Brain Health Longitudinal Study. Baseline micro- and macro-cerebrovascular abnormalities were evaluated by MRI brain on recruitment and received COVID-19 vaccination (SinoVac or BioNTech).
  Interventions: Diagnostic Test: Laboratory tests and Montreal Cognitive Assessment
- Control Group: Citizens who received baseline cognitive assessment and evaluation of metabolic risk factors from the CUHK Brain Health Longitudinal Study. Baseline micro- and macro-cerebrovascular abnormalities were evaluated by MRI brain on recruitment and have not received any COVID-19 vaccines nor clinically/serologically evident SARS-CoV-2 infection.
  Interventions: Diagnostic Test: Laboratory tests and Montreal Cognitive Assessment

INTERVENTIONS:
Diagnostic Test: Laboratory tests and Montreal Cognitive Assessment — Laboratory tests at baseline and 16 weeks (+/-4 weeks) after 2nd dose of vaccine and serological testing for IgG antibody. Participants who have a scheduled vaccination date shall undergo an MRI brain 16 weeks (+/-4 weeks) after the second dose of COVID-19 vaccination (either SinoVac or BioNTech). A face-to-face assessment 16 weeks (+/-4 weeks) will also be conducted after the 2nd dose of COVID-vaccine for evaluation of any clinical events, followed by a phone visit every 6 months. Cognitive assessment by MoCA will be performed at baseline, 16 weeks (+/-4 weeks) then every 12 months after the 2nd dose of COVID-19 vaccine.
  Groups: Vaccination Group
Diagnostic Test: Laboratory tests and Montreal Cognitive Assessment — Laboratory tests at baseline and serological testing for IgG antibody to exclude past COVID-19 infection. The timing of the second MRI brain, laboratory tests, clinical and cognitive assessment will be matched with the timing in the vaccination group are available.
  Groups: Control Group

SUMMARY:
Safe and effective severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccines may reduce the transmission of and achieve population immunity against the COVID-19 pandemic, which accounted for more than 3.75million deaths worldwide. With World Health Organization's (WHO) effort on ensuring equitable access to COVID-19 vaccines, vaccination rate may increase in the near future.

On the other hand, vaccination hesitancy has emerged as a major hindrance on the global vaccination campaigns in certain areas due to safety concerns, social factors, and public health policies. For instance, a recent survey conducted in Hong Kong showed a low vaccine acceptance rate of 37%. Long-term safety concerns and post-vaccination events relayed by the social media maybe reasons for vaccination hesitancy. Among which, cerebrovascular accidents (CVA) after vaccination were one of the most frequently reported post-vaccination events. These reports ranged from ischemic strokes in elderly patients with multiple cardiovascular co-morbidities, to hemorrhage strokes in otherwise "young-and-fit" adults. While many of these events were investigated by the COVID-19 immunization expert committee, an important premise to address the apprehension of CVA after vaccination is the provision of evidence-based information of the impact of COVID-19 vaccines on brain health.

In this prospective, longitudinal, observational study, we aim to elucidate the relationship between COVID-19 vaccines and cerebrovascular health in healthy citizens in a population-based cohort.

DETAILED DESCRIPTION:
We shall recruit all consecutive citizens from a prospective, population-based cohort from the CUHK Brain Health Longitudinal Study free of clinically evident neurological diseases. The CUHK Brain Health Longitudinal Study cohort comprises of an epidemiologically representative sample from all socio-economic classes in the 18 districts of Hong Kong with reference to government census data. All citizens received baseline cognitive assessment and evaluation of metabolic risk factors. Baseline micro- and macro-cerebrovascular abnormalities were evaluated by MRI brain on recruitment.

We shall phone contact the citizens who met the inclusion criteria to enquire their vaccination plan. Citizens who received COVID-19 vaccination (SinoVac or BioNTech) and willing to join the study, our services coordinator, co-investigator or principal investigator will interview and explain the study in details and obtain the participant's consent. After signing the consent, the participant shall undergo a 2nd MRI brain 16 weeks (+/-4 weeks) after the 2nd dose of vaccination. The control group is defined as citizens who have not received any COVID-19 vaccines nor clinically/serologically evident SARS-CoV-2 infection.

We shall collect the following information for the vaccination group:

Demographic data ; Medical co-morbidities ; Laboratory tests at baseline and 16 weeks (+/-4 weeks) after 2nd dose of vaccine and serological testing for IgG antibody. We shall conduct a face-to-face assessment 16 weeks (+/-4 weeks) after the 2nd dose of COVID-vaccine for evaluation of any clinical events, followed by a phone visit every 6 months. Cognitive assessment by MoCA will be performed at baseline, 16 weeks (+/-4 weeks) then every 12 months after the 2nd dose of COVID-19 vaccine.

On the other hand, we shall collect the following information for the control group:

Demographic data ; Medical co-morbidities ; Laboratory tests at baseline and serological testing for Immunoglobulin G (IgG) antibody to exclude past COVID-19 infection prior to the second MRI brain.The timing of the second MRI brain, laboratory tests, clinical and cognitive assessment in the control group will be matched with the timing in the vaccination group are available.

The proposed study does not involve formulating new diagnoses or directly offering treatment for neurological and/or psychiatric conditions. All patients admitted to PWH or other medical institutes will be treated according to the standard care at the corresponding institution, regardless of their decision to participate in this repository. Should results from this study lead to discovery of one or more factors associated with development of brain disease, the principal investigators, co-investigators, or study coordinator will inform, counsel and offer diagnostic and/or therapeutic recommendations to participants accordingly. The participants may be referred to relevant departments for follow-up clinical visits.

Safe and effective SARS-CoV-2 vaccines may reduce the transmission of and achieve population immunity against the COVID-19 pandemic, which accounted for more than 3.75million deaths worldwide. However, vaccination hesitancy has emerged as a major hindrance on the global vaccination campaigns in certain areas due to safety concerns, social factors, and public health policies. The proposed study will allow us to address the apprehension of cerebrovascular accidents after vaccination is the provision of evidence-based information of the impact of COVID-19 vaccines on brain health.

ELIGIBILITY:
Inclusion Criteria:

All consecutive citizens in the CUHK Brain Health Longitudinal Study cohort who received baseline MRI brain.

Exclusion Criteria:

1. Citizens with clinically evident stroke or dementia prior to recruitment; or
2. Citizens who are unable to provide an informed consent; or
3. Citizen with contraindications to MRI brain, e.g., non-MRI compatible implants, claustrophobia, etc; or
4. Citizens who had no baseline MRI brain assessment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Chinese ONLY 2. Hong Kong Resident
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-07-05 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Imaging markers | December, 2026
  We shall perform cranial MRI examinations in a 3-Tesla scanner (MAGNETOM Prisma; Siemens AG, Munich, Germany). The scanning protocol will employ a standard stroke protocol MRI scan with axial T1-weighted, T2-weighted, FLAIR, susceptibility weighted imaging, diffusion weighted imaging, and time-of-flight magnetic resonance angiography (MRA) sequences.
Imaging analysis | December, 2026
  Blinded to the time sequence, clinical outcomes and the vaccination status, an experienced neuro-radiologist and an experienced stroke neurologist shall independently evaluate the imaging markers (as stated in endpoint assessment above). Disparity will be resolved by discussion. White matter hyperintensity volume will be gauged by FMRIB's Software Library Brain Intensity Abnormality Classification Algorithm (BIANCA), a fully automated, supervised method for white matter hyperintensities detection. Brain volume will be measured by FMRIB's Software Library voxel-based morphometry analysis.Siemens AG, Munich, Germany). The scanning protocol will employ a standard stroke protocol MRI scan with axial T1-weighted, T2-weighted, FLAIR, susceptibility weighted imaging, diffusion weighted imaging, and time-of-flight magnetic resonance angiography (MRA) sequences.

CONTACTS AND LOCATIONS:
Overall Officials: Bonaventure Yiu Ming IP, MB ChB, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No